CLINICAL TRIAL: NCT04861623
Title: A Pilot Clinical Trial to Assess the Effects of 100% Orange Juice on Skin Health in Women Using a Randomized Double-Blinded Placebo-Controlled Crossover Design
Brief Title: Effects of 100% Orange Juice on Skin Health in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB202100814
Record Dates: First submitted 2021-04-20; First posted 2021-04-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-03

CONDITIONS: Skin Health
Keywords: Orange Juice; Skin health

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the identity of the beverages
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orange Juice then Placebo juice (SunnyD) (Active Comparator): Participants will be provided orange juice for 84 days in this arm. After 28 days wash-out period, participants will receive Fanta for 84 days.
  Interventions: Other: Orange juice; Other: Placebo juice (SunnyD)
- Placebo (SunnyD) then Orange juice (Active Comparator): Participants will be provided Fanta for 84 days in this arm. After 28 days wash-out period, participants will receive Orange juice for 84 days.
  Interventions: Other: Orange juice; Other: Placebo juice (SunnyD)

INTERVENTIONS:
Other: Orange juice — Orange juice will be purchased commercially.
Other: Placebo juice (SunnyD) — SunnyD beverage will be purchased commercially.

SUMMARY:
Daily consumption of Orange Juice (OJ) protects skin against UV-induced damages and wrinkling, improves skin barrier function and overall skin health by decreasing oxidative stress, inflammation, and protein glycation. The positive effects of OJ on skin appearance are associated with improvements of the stratum corneum lipidomic and skin microbiome.

DETAILED DESCRIPTION:
There is a lack of clinical evidence on how 100% orange juice (OJ) affects skin health. Women make over 90% of the decisions on food purchases for family. Skin health is a major concern for women because skin ageing becomes visibly noticeable after age 30 due to UV exposure, oxidative stress, and collagen glycation. The investigators hypothesize that micronutrients in OJ, including vitamin C, flavanones, and carotenoids, protect skin against photoaging and wrinkling by alleviating oxidative stress, inflammation, and collagen glycation. The investigators further propose that daily OJ consumption (16 oz) will improve skin elasticity, barrier function, overall skin appearance and health. The study hypotheses will be tested in a 12-week clinical trial in 24 women aged 45-65 using a randomized, double-blinded, placebo-controlled, crossover design. Placebo will be formulated using SunnyD orange-flavered beverage to match the color, taste, and calorie content of OJ. This research will measure UV-induced skin erythema, wrinkles, smoothness, roughness, elasticity, hydration, pH, melanin, and transepidermal water loss (a skin barrier index) of skin on both face and forearm. Skin strips and swabs will be collected and preserved for future assessments of skin lipids and colonized microorganisms (skin microbiome) because they are key factors affecting skin health. Positive results from this pilot trial will provide clinical evidence on the effectiveness of OJ to maintain skin health and reduce ageing. This research will be carried out by a research team with the experience and facilities for skin research.

ELIGIBILITY:
Inclusion Criteria:

* BMI (18.5-29.9)
* Body weight ≥110 pounds
* Fitzpatrick skin type 2 and 3.

Exclusion Criteria:

* pregnancy
* breast-feeding
* impaired fasting glucose
* frequent alcohol use
* history of skin cancer
* sunbathing and the use of tanning bed, intake of vitamin/mineral supplements
* habitual high intake of fruits (≥ 2 cups daily)
* intake of medication that might influence the outcome of the study

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Skin UV sensitivity | Baseline, 84 days
  Irradiation will be applied to dorsal skin (back, scapular region not typically exposed to the sun) with 2 times of minimal erythema dose using an FDA approved UVB phototherapy light and a UV light meter. At baseline, after 42 and 84 days, skin color will be measured before and 24 hours after irradiation. Skin color will be evaluated by a colorimeter. The a*-value (red/green-axis) is a measure of reddening (erythema).

SECONDARY OUTCOMES:
Skin transepidermal water loss | Baseline, 84 days
  Skin transepidermal water loss will be measured using a Tewameter to evaluate the water barrier function of the skin.
Skin erythema and melanin index | Baseline, 84 days
  Skin erythema and melanin index will be assessed with Mexameter. These two components are mainly responsible for the color of the skin. They are measured by reflectance.
Inflammation biomarkers | Baseline, 84 days
  Plasma levels of C-reactive proteins will be analyzed as inflammation biomarkers using ELISA kits.
Inflammation biomarkers | Baseline, 84 days
  Plasma levels of IL-6 proteins will be analyzed as inflammation biomarkers using ELISA kits.
oxidative stress | Baseline, 84 days
  Malondialdehyde in plasma will be determined as a marker of lipid peroxidation using a photometric method.
skin hydration | Baseline, 84 days
  Skin hydration will be measured using a Skin Corneometer.
skin pH | Baseline, 84 days
  Skin pH will be measured using a Skin-pH-Meter.

CONTACTS AND LOCATIONS:
Locations (1):
- Food Science and Human Nutrition Department at University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Li R, Kim MH, Sandhu AK, Gao C, Gu L. Muscadine Grape (Vitis rotundifolia) or Wine Phytochemicals Reduce Intestinal Inflammation in Mice with Dextran Sulfate Sodium-Induced Colitis. J Agric Food Chem. 2017 Feb 1;65(4):769-776. doi: 10.1021/acs.jafc.6b03806. Epub 2017 Jan 23. PMID 28112913
- [Background] Heinrich U, Moore CE, De Spirt S, Tronnier H, Stahl W. Green tea polyphenols provide photoprotection, increase microcirculation, and modulate skin properties of women. J Nutr. 2011 Jun;141(6):1202-8. doi: 10.3945/jn.110.136465. Epub 2011 Apr 27. PMID 21525260
- [Background] Heinrich U, Neukam K, Tronnier H, Sies H, Stahl W. Long-term ingestion of high flavanol cocoa provides photoprotection against UV-induced erythema and improves skin condition in women. J Nutr. 2006 Jun;136(6):1565-9. doi: 10.1093/jn/136.6.1565. PMID 16702322
- [Background] Heckman CJ, Chandler R, Kloss JD, Benson A, Rooney D, Munshi T, Darlow SD, Perlis C, Manne SL, Oslin DW. Minimal Erythema Dose (MED) testing. J Vis Exp. 2013 May 28;(75):e50175. doi: 10.3791/50175. PMID 23748556
- [Background] Manippa V, Padulo C, van der Laan LN, Brancucci A. Gender Differences in Food Choice: Effects of Superior Temporal Sulcus Stimulation. Front Hum Neurosci. 2017 Dec 7;11:597. doi: 10.3389/fnhum.2017.00597. eCollection 2017. PMID 29270120